CLINICAL TRIAL: NCT01742390
Title: A Multicenter Study to Evaluate the Effects of Switching to Aripiprazole 12 Weeks on the Sexual Dysfunction From Risperidone or Paliperidone in Patients With Schizophrenia Spectrum Disorders or Bipolar Spectrum Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Si Tianmei (Other)
Responsible Party: Sponsor-Investigator, Si Tianmei, Professor, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARI_IIT_01/02
Record Dates: First submitted 2012-11-22; First posted 2012-12-05 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Sexual Dysfunction; Hyperprolactinemia
Keywords: schizophrenia; risperidone; paliperidone; aripiprazole
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Hyperprolactinemia; Schizophrenia | interventions — Aripiprazole; Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Experimental): Plateau switch to aripiprazole (ARI) from risperidone (RIS) or paliperidone (PALI)
  Interventions: Drug: Aripiprazole
- risperidone or paliperidone (Active Comparator): Stay on risperidone (RIS) or paliperidone (PALI)
  Interventions: Drug: risperidone or paliperidone

INTERVENTIONS:
Drug: Aripiprazole — Plateau switch to aripiprazole (ARI) from risperidone (RIS) or paliperidone (PALI)
  Arms: Aripiprazole
Drug: risperidone or paliperidone
  Arms: risperidone or paliperidone

SUMMARY:
This trial designed to investigate the effect of switching to aripiprazole from risperidone or paliperidone on reverse prolactin level, and consequently improve sexual dysfunction in adult patients with schizophrenia spectrum disorders and bipolar spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12-55 years (male), 12-40 (female)
2. Diagnosis: Schizophrenia spectrum disorders & bipolar spectrum disorders (only Korea) by DSM-IV-TR
3. Receiving RIS or PALI with stable dose for > 1 month by their physician;
4. Prolactin level Adult: > 20 ng/ml (male), 25 ng/ml (female) Child/Adolescent: > 20 ng/ml (male, female)
5. Children and adolescents (age: 12~17 years) having more than one sexual system dysfunction measured by 5 of the 48 UKU items (galactorrhoea, gynecomastia and erectile dysfunction for male, galactorrhea, amenorrhoea/oligomenorrhoea, and dry vagina for female) or Adults (age: 18~55 years) who are considered to have sexual/reproductive dysfunction if they had either a total score of 19 or higher; a score of 5 or higher on one question; or a score of 4 or higher on 3 questions.
6. Subjects who have consented to participate by signing an informed consent form.

   -

Exclusion Criteria:

1. Medical disorder or psychiatric comorbidity or condition known to affect prolactin, sex hormone balance or bone metabolism (i.e., unstable medical disease, Cushing's disease, chronic renal failure, thyroid dysfunction, eating disorder)
2. History of hematological and/or solid malignancies
3. Physical or functional obstruction to food intake or impaired digestive/absorptive function
4. Known hypersensitivity to any study medication (risperidone, paliperidone, and aripiprazole)
5. Insulin requiring diabetes mellitus or poorly controlled diabetes mellitus (HbA1c > 9% or change of antidiabetics treatment within the 12weeks prior to screening)
6. Uncontrolled hypertension (SBP/DBP 140/90 mmHg), congestive heart failure (NYHA class III or IV), other significant cardiovascular illness (myocardial infarction, unstable angina, cardiac arrhythmia etc.)
7. Baseline QTc interval of > 450 msec
8. Hepatic and/or renal dysfunction

1) Bilirubin level ≥ 1.5 upper normal limits 2) AST/ALT ≥ 3 UNL or 3) Serum creatinine ≥ 1.5 9. Any patient hospitalized for acute exacerbation of their condition within 2 months of randomization 10. Recent (within the past 1 month) or planned treatment with prohibited medications in the protocol

-

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in severity of sexual/reproductive system dysfunction at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Percentage of absence of sexual/reproductive system dysfunction on the UKU side effect rating scale or ASEX | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Institute of mental health, Peking University, Beijing, Beijing Municipality
  - The first hospital of Hebei Province University, Shijiazhuang, Hebei